CLINICAL TRIAL: NCT02763592
Title: Impact of 5% Lidocaine Medicated Plaster on Allodynic Symptoms of Localized Neuropathic Pain After Knee Surgery
Acronym: LiNe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0261; RBHP 2015 PICKERING 4 (Other: CHU Clermont-Ferrand)
Record Dates: First submitted 2016-04-11; First posted 2016-05-05 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Allodynic Symptoms; Localized Neuropathic Pain
Keywords: Localized Neuropathic pain; 5% lidocaine medicated plaster; Knee surgery
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lidocaine (Experimental): This is a randomized, placebo-controlled, double-blind, parallel-group clinical trial comparing 5% lidocaine medicated plaster (5LP) and placebo whether neuropathic pain symptoms (dynamic mechanical allodynia, pressure, hot and cold) have a different chronological improvement with 5LP compared to placebo
  Interventions: Drug: Lidocaine
- placebo (Placebo Comparator): This is a randomized, placebo-controlled, double-blind, parallel-group clinical trial comparing 5% lidocaine medicated plaster (5LP) and placebo whether neuropathic pain symptoms (dynamic mechanical allodynia, pressure, hot and cold) have a different chronological improvement with 5LP compared to placebo
  Interventions: Other: placebo plaster

INTERVENTIONS:
Drug: Lidocaine — The aim of this study is to evaluate the impact of 5% lidocaine medicated plaster on allodynic symptoms of localized neuropathic pain after knee surgery
  Arms: Lidocaine
Other: placebo plaster — This is a randomized, placebo-controlled, double-blind, parallel-group clinical trial comparing 5% lidocaine medicated plaster (5LP) and placebo whether neuropathic pain symptoms (dynamic mechanical allodynia, pressure, hot and cold) have a different chronological improvement with 5LP compared to placebo. Pain intensity and pain relief, sleep and quality of life and osteoarthritis severity are also assessed.
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the impact of 5% lidocaine medicated plaster on allodynic symptoms of localized neuropathic pain after knee surgery.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, parallel-group clinical trial comparing 5% lidocaine medicated plaster (5LP) and placebo whether neuropathic pain symptoms (dynamic mechanical allodynia, pressure, hot and cold) have a different chronological improvement with 5LP compared to placebo. Pain intensity and pain relief, sleep and quality of life and osteoarthritis severity are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 80 years
* Male or female, for women of childbearing potential, a negative pregnancy test
* Patients with PONP following knee surgery
* Patients with neuropathic pain DN4 ≥ 4
* Patients at least 3 months post-surgery
* Patients suffering from at least the allodynic brush-induced mechanical allodynia symptom (DMA) rated as ≥ 5/10 on the numerical scale
* Patient with no localized neuropathic pain symptoms (DN4<4) on the contralateral knee
* Intact skin besides the scar of surgery (absence of skin disease, skin irritation, inflammation or injury, such as active herpes zoster lesions, atopic dermatitis, wounds) in the area where the medicated plasters will be applied
* Naive from Versatis® treatment
* Treated with stable systemic analgesic and planned to remain stable all over the duration of the study
* Insured by French social security
* Included or agreement to be included in the national register of participants in biomedical research

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time to response to treatment | from inclusion to 3 months
  Time to response to treatment defined as a 30% reduction in dynamic brush-induced mechanical allodynia on the localized pain area during the chronological period extending from inclusion to 3 months

SECONDARY OUTCOMES:
- Kinetics of evolution over time of pain evaluated by numeric scale ranging from 0 to 10 with brush-induced Dynamic Mechanical Allodynia (DMA) in both groups (Placebo and 5LP) | from inclusion to 3 months
  Kinetics of evolution over time of pain evaluated by numeric scale ranging from 0 to 10 with brush-induced Dynamic Mechanical Allodynia (DMA) in both groups (Placebo and 5LP)
- Kinetics of evolution over time of pain evaluated by numeric scale ranging from 0 to 10 with Mechanical Detection Threshold (MDT) in both groups (Placebo and 5LP) | at inclusion
  - Kinetics of evolution over time of pain evaluated by numeric scale ranging from 0 to 10 with Mechanical Detection Threshold (MDT) in both groups (Placebo and 5LP)
- Kinetics of evolution over time of Cold Detection Threshold (CDT) and Warm Detection Threshold (WDT) in both groups (Placebo and 5LP) | at inclusion
  - Kinetics of evolution over time of Cold Detection Threshold (CDT) and Warm Detection Threshold (WDT) in both groups (Placebo and 5LP)
Pain evaluated with numerical rating scale ranging from 0 to 10 | at inclusion
  Pain evaluated with numerical rating scale ranging from 0 to 10
Pathophysiology of neuropathic characteristics with DN4 questionnaire | at inclusion
  Pathophysiology of neuropathic characteristics with DN4 questionnaire
Evolution of the size of the allodynic area | at inclusion
- Responder rate, defined as 30% and 50% reduction over time on pain evaluated by numeric scale ranging from 0 to 10 with brush-induced Dynamic Mechanical Allodynia (DMA) | at 3 months
  - Responder rate, defined as 30% and 50% reduction over time on pain evaluated by numeric scale ranging from 0 to 10 with brush-induced Dynamic Mechanical Allodynia (DMA)
- Responder rate, defined as 30% and 50% reduction over time on pain evaluated by numeric scale ranging from 0 to 10 with Mechanical Detection Threshold (MDT) | at 3 months
  - Responder rate, defined as 30% and 50% reduction over time on pain evaluated by numeric scale ranging from 0 to 10 with Mechanical Detection Threshold (MDT)
- Responder rate, defined as 30% and 50% reduction over time on Cold Detection Threshold (CDT) and Warm Detection Threshold (WDT) | at 3 months
  - Responder rate, defined as 30% and 50% reduction over time on Cold Detection Threshold (CDT) and Warm Detection Threshold (WDT)
- Comparison of pain evaluated by numeric scale ranging from 0 to 10 with brush-induced Dynamic Mechanical Allodynia (DMA) between painful knee and contralateral knee on the same anatomic location. | at 3 months
  - Comparison of pain evaluated by numeric scale ranging from 0 to 10 with brush-induced Dynamic Mechanical Allodynia (DMA) between painful knee and contralateral knee on the same anatomic location.
- Comparison of pain evaluated by numeric scale ranging from 0 to 10 with Mechanical Detection Threshold (MDT) between painful knee and contralateral knee on the same anatomic location | at 3 months
  - Comparison of pain evaluated by numeric scale ranging from 0 to 10 with Mechanical Detection Threshold (MDT) between painful knee and contralateral knee on the same anatomic location
- Comparison of Cold Detection Threshold (CDT) and Warm Detection Threshold (WDT) between painful knee and contralateral knee on the same anatomic location. | at 3 months
  - Comparison of Cold Detection Threshold (CDT) and Warm Detection Threshold (WDT) between painful knee and contralateral knee on the same anatomic location.
Evolution of sleep by Pittsburgh Sleep Quality Index (PGIC) questionnaire. | at 3 months
  Evolution of sleep by Pittsburgh Sleep Quality Index (PGIC) questionnaire.
Evolution of quality of life by Short-Form 12 (SF-12) questionnaire. | at 3 months
  Evolution of quality of life by Short-Form 12 (SF-12) questionnaire.
Evolution of Patient Global Impression of Change (PGIC) questionnaire | at 3 months
  Evolution of Patient Global Impression of Change (PGIC) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pickering G, Voute M, Macian N, Ganry H, Pereira B. Effectiveness and safety of 5% lidocaine-medicated plaster on localized neuropathic pain after knee surgery: a randomized, double-blind controlled trial. Pain. 2019 May;160(5):1186-1195. doi: 10.1097/j.pain.0000000000001502. PMID 31009419